CLINICAL TRIAL: NCT01891591
Title: Assessment of Nutritional Status and Vitamin Deficiencies in Obese Subjects After Gastric Bypass Surgery
Brief Title: Assessment of Nutritional Status After Gastric Bypass Surgery
Status: Completed | Type: Observational
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Luc Tappy, MD, professor of Physiology, University of Lausanne
Other Study IDs: 39/08
Record Dates: First submitted 2013-06-17; First posted 2013-07-03 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-06

CONDITIONS: Obesity; Nutritional Deficiencies
Keywords: Obesity; Gastric bypass; Energy balance; Nutritional status; Protein balance
MeSH Terms: conditions — Obesity; Malnutrition | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- obese female subjects: 16 obese female subjects with BMI > 40 kg/m2 on a waiting list for bariatric surgery
  Interventions: Procedure: Roux-en-Y gastric bypass (RYGP)

INTERVENTIONS:
Procedure: Roux-en-Y gastric bypass (RYGP)

SUMMARY:
This study is aimed at assessing how Roux-en-Y gastric bypass (RYGP) impacts on energy and nutrients' intake, energy expenditure, and nutritional status in obese patients. It will try quantitate energy and protein balance after RYGP, and to identify how RYGP effects the intake of various common dietary protein sources 16 female patients with BMI > 40 kg/m2 and on a waiting list for bariatric surgery will be included. The following measurements will be performed before, and 1, 3, 6, 12, and 36 months after RYGP

* body weight
* body composition (bio impedancemetry)
* basal metabolic rate (open circuit indirect calorimetry)
* 24-hour urinary urea excretion
* fasting blood chemistry
* energy and macronutrient's intake (3-day dietary recall)

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* gender: females
* body mass index >35 kg/m2

Exclusion Criteria:

* GI tract diseases
* endocrine diseases

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 16 female obese subjects on a waiting list for gastric bypass bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2008-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
changes in daily dietary protein intake | measurements obtained baseline , and 1,3, 6, 12, 36 months after surgery
  changes in 24-hour protein intake will be evaluated by 7-day food diary; portion size will be assessed with the use of photographs from the SU.VI.MAX study

SECONDARY OUTCOMES:
changes in total energy intake | measurements obtained baseline , and 1,3, 6, 12, 36 months after surgery
  changes in 24-hour energy intake will be evaluated by 7-day food diary; portion size will be assessed with the use of photographs from the SU.VI.MAX study
changes in basal metabolic rate | measurements obtained baseline , and 3, 6, 12, 36 months after surgery
  BMR will be measured by indirect calorimetry over a 45-90 min period
changes in total energy intake | measurements obtained baseline , and 1,3, 6, 12, 36 months after surgery
  Changes in daily total energy intake will be evaluated by 7-day food diary; portion size will be assessed with the use of photographs from the SU.VI.MAX study

OTHER OUTCOMES:
changes in fasting, resting respiratory exchange ratio | measurements obtained baseline, and 3, 6, 12, and 36 months after RYGP
  measurement will be obtained by indirect calorimetry
changes in 24-hour urinary urea excretion | Measurements obtained baseline , and 3, 6, 12, 36 months after RYGP
  24-hour urine collections

CONTACTS AND LOCATIONS:
Overall Officials: Vittorio Giusti, MD, Principal Investigator — CHUV
Locations (1):
- Clinical Research Centre, CHUV, Lausanne, Switzerland

REFERENCES:
- [Derived] Chakhtoura MT, Nakhoul NF, Akl EA, Safadi BY, Mantzoros CS, Metzendorf MI, El-Hajj Fuleihan G. Oral vitamin D supplementation for adults with obesity undergoing bariatric surgery. Cochrane Database Syst Rev. 2024 Oct 1;10(10):CD011800. doi: 10.1002/14651858.CD011800.pub2. PMID 39351881
- [Derived] Giusti V, Theytaz F, Di Vetta V, Clarisse M, Suter M, Tappy L. Energy and macronutrient intake after gastric bypass for morbid obesity: a 3-y observational study focused on protein consumption. Am J Clin Nutr. 2016 Jan;103(1):18-24. doi: 10.3945/ajcn.115.111732. Epub 2015 Dec 16. PMID 26675775
- [Derived] De Giorgi S, Campos V, Egli L, Toepel U, Carrel G, Cariou B, Rainteau D, Schneiter P, Tappy L, Giusti V. Long-term effects of Roux-en-Y gastric bypass on postprandial plasma lipid and bile acids kinetics in female non diabetic subjects: A cross-sectional pilot study. Clin Nutr. 2015 Oct;34(5):911-7. doi: 10.1016/j.clnu.2014.09.018. Epub 2014 Sep 26. PMID 25306425